CLINICAL TRIAL: NCT05355831
Title: Patient-tailored Transcranial Direct Current Stimulation to Improve Stroke Rehabilitation
Acronym: PRACTISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christina Kruuse (Other)
Collaborators: Danish Research Centre for Magnetic Resonance (Other); The Novo Nordic Foundation (Other); University of Copenhagen (Other); Lundbeck Foundation (Other)
Responsible Party: Sponsor-Investigator, Christina Kruuse, Study Principal Investigator, Consultant Neurologist, Dept. Neurology, Herlev Hospital, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H-20036199
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke; Upper Extremity Hemiparesis
Keywords: non-invasive brain stimulation; transcranial direct current stimulation; effective connectivity; functional connectivity; Fugl-Meyer Assessment; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Intervention pilot- and feasibility trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Transcranial Direct Current Stimulation (Active Comparator): Anodal TDCS 1mV for 2x 20 minutes.
  Interventions: Device: Active Transcranial Direct Current Stimulation
- Sham stimulation (Sham Comparator): 2x 20 minutes of sham stimulation (30 sec ramp up, followed by current of 0 for 18.5 minutes followed by 30 sec ramp down).
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation — See arm/group description
  Arms: Active Transcranial Direct Current Stimulation
Device: Sham stimulation — See arm/group description
  Arms: Sham stimulation

SUMMARY:
In a double-blinded sham-controlled study the effect of patient-tailored transcranial direct current stimulation during rehabilitation training will be examined.

DETAILED DESCRIPTION:
Approximately two thirds of stroke patients have reduced motor function which have a large impact on both activities of daily living and quality of life. Only 12-34% achieve full motor recovery.

There is a growing interest in using non-invasive brain stimulation (NIBS) techniques to supplement neurorehabilitation. NIBS can modulate cortical excitability and is a powerful tool for motor rehabilitation post-stroke. Application Transcranial Direct Current Stimulation (TDCS) is currently emerging as a tool used in neurorehabilitaiton. Prior studies have shown that TDCS-stimulation prior to physical training may significantly improve of motor function post-stroke. However, up to 50% of the participants recieving active TDCS show no response to stimulation.

A one-size-fits-all approach to TDCS in stroke rehabilitation may not be optimal and a more precise and individualized targeting is warranted to stimulate functionally relevant areas.

In this study TDCS will be personalized for stroke patients with upper-extremity paresis using individual functional and structural Magnetic Resonance Imaging (MRI) and an electric field modelling pipeline developed at Danish Research Centre for Magnetic Resonance (DRMCR). Based on these measures the electric current induced by TDCS will individually target the area with residual neural activity during movement. The effect of personalized TDCS will be assessed by clinical measures of motor improvement. Sub-studies furthermore assess if the functional reorganization of motor networks is affected by personalized TDCS by application of functional magnetic resonance (fMRI) and.

The study will have 3 phases:

1. Personalization: The stimulation profile of each patient will be individualized using structural MRI a pipeline for simulation based on MRI (SimNIBS) to make individual anatomical head models in order to estimate the best montage and current dosage. Further, task-based fMRI will be used to estimate residual motor activity location. The target current is set in the area displaying the highest residual motor activity in sensorimotor areas.
2. Intervention: Four weeks upper extremity training program of specialized supervised physiotherapeutic training 3 times per week. Each training session consists of 2x 20 minutes of training with concurrent personalized TDCS stimulation or montage of equipment but no stimulation (sham). Each bloc of 20 minutes training is separated by a small break of 5-10 minutes. Both patient, therapist and investigator will be blinded to the stimulation mode (activ TDCS or sham)
3. Follow-up: Immediately after the 4 weeks of intervention and 12 weeks after intervention has ended, follow-up with clinical examination and brain MRI will be done.

Ad baseline Transcranial Magnetic Stimulation (TMS) will be done as well to assess corticospinal integrity as well as estimation of intracortical inhibition.

Hypothesis:

The main hypothesis is that personalized ipsi-lesional anodal TDCS during specialized individualized arm-training will lead to significantly greater improvements in upper-extremity motor function compared to sham.

Substudy with healthy controls:

A cohort of 20 healthy age- and sex matched controls will be recruited for one session of MRI and TMS identical to the procedure of the patients at baseline as well as the same questionnaires (Protocol amendment approved by the local Ethics Committee the 10th October 2022).

These data will be analyzed in a substudy for normative comparison between the stroke patients and healthy age- and sex-matched controls.

Hypothesis - Healthy Controls:

Stroke patients will exhibit a higher laterality index measured by fMRI and a stronger degree of interhemispheric inhibition at baseline compared to healthy controls measued by task-related fMRI and by TMS iSP and SICI.

The degree of interhemispheric inhibition in stroke patients will normalize during recovery and be similar to normal controls at the last follow-up after 12 weeks.

Further, the degree of normalization of the interhemispheric inhibition in stroke patients will be proportional to degree of improvement of the upper-extremity measured by UE-FMA.

July 2024:

Due to challenging recruitment and at much lower recruitment rate than expected the trial design was changed from superiority to pilot- and feasibility trial. Therefore, the sample size was correspondingly adjusted to expected 24 with 12 participants in each of the two arms. Furthermore, outcome measures were re-prioritized to also contain feasibility outcome measures and primary outcome was changed to follow-up Fugl-Meyer Assessment score of upper-extremity (FMA-UE) adjusted for baseline in stead of change in FMA-UE from baseline to follow-up.

ELIGIBILITY:
Patients - Inclusion Criteria:

1. Age >18 years
2. Ischemic stroke confirmed by clinical and imaging criteria
3. Hemiparesis including reduced upper-extremity function
4. Location of stroke either cortically involving middle cerebral artery or the anterior cerebral artery circulation or subcortical (involving thalamus, basal ganglia).
5. NIHSS score >2 and <8
6. Modified Rankin Scale (mRS) ≤ 3
7. Index of stroke within 4 weeks of inclusion
8. Signed informed consent

Patients - Exclusion Criteria:

1. >50% stenosis of extra- or intracranial artery as well as vascular malformations or aneurisms detected by brain CT-angiography.
2. Exclusively ischemic stroke in spine, pons, brainstem, medulla or cerebellum.
3. History of seizures, epilepsy, anxiety, dementia alcohol- or drug abuse.
4. Prior serious head injury or neurosurgery
5. Frequent severe headaches or migraine.
6. Pregnancy or breastfeeding
7. Current use of neuro-receptor/transmitter modulating medication, or medication interfering with seizure threshold (such as antiepileptic medication, some antidepressants, anxiety medication, antihistamines, stimulant drugs for attention deficit hyperactivity disorder).
8. Pacemaker, implantable cardiac device unit (ICD-unit), metal fragments or other materials implanted not compatible with MRI (see appendix B).
9. Claustrophobia
10. Prior adverse effect to TDCS or Transcranial Magnetic Stimulation.
11. Not able to provide informed consent.
12. Terminally ill or short life expectancy.

Healthy controls - Inclusion criteria:

1. Age between >18 years (matched to patients)
2. Sex and age matched to patients
3. Able bodied
4. Have the ability to comply with all requirements of the study protocol, as determined by the investigator
5. No history of stroke or dementia
6. Eligible for MRI and TMS

Healthy controls - Exclusion Criteria:

1. History of neurologic disease
2. History of cerebral haemorrhage or brain damage
3. Pregnancy
4. Pacemaker or other implanted electronic devices
5. Claustrophobia
6. Psychiatric disorder
7. Epilepsy or close relatives suffering from epilepsy
8. Migraine
9. Any contraindication to MRI or TMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-08-28 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pilot outcome | From baseline to four months
  Difference in Upper-extremity Fugl-Meyer Assessment (UE-FMA) score at end of treatment. Range 0-66.

SECONDARY OUTCOMES:
Change in upper-extremity function | From baseline to four months
  Difference in change in Action Reach Arm Test (ARAT) score. Range 0-57. High scores mean a better outcome.
Stroke severity | From baseline to four months
  Difference in change in National Health Institutes Stroke Scale (NIHSS). Range 0-42. High scores mean a better outcome.
Stroke disability | From baseline to four months
  Difference in change in Modified Rankin Scale (mRS). Range 0-6. Lower scores mean a better outcome.
ADL performance | From baseline to four months
  Difference in change in Bartel's 20-item Index (BI-20). Range 0-100. Higher scores mean better outcome.
Gait speed | From baseline to four months
  Difference in change in 10 Meter Walk Test (10MWT) in minutes:sec.
Physical Activity | From baseline to four months
  Difference in change in Physical Activity Scale 2.0 (PAS2). The answers will be translated into a Metabolic Equivalent of Task (MET)-score. The higher MET-score the higher level of activity.
Montreal Cognitive Assessment | From baseline to four months
  Difference in change in Montreal Cognitive Assessment (MoCA) score. Score range 0-30. Higher scores mean a better outcome.
Symbol Digit Modalities Test | From baseline to four months
  Difference in change in Symbol Digit Modalities Test (SDMT) score. Score range 0-110. Higher scores mean a better outcome.
Health-related quality of life | From baseline to four months
  Difference in change in EQ-5D-5L score. Range 1 to 20, a high score means low health-related quality of life. Includes a 0-100 visual analogue scale for overall percieved quality of life.
Becks Depression Inventory (BDI) | From baseline to four months
  Difference in change in BDI-II score. Score range 0-63. Higher score means increased risk of depression.
Fatigue Severity Scale (FSS) | From baseline to four months
  Difference in change in FSS score. Score range 0-7. Higher score means increased fatigue severity.
WHO-5 Well-Beeing Index | From baseline to four months
  Difference in change in WHO-5 score. Score range 0-100. Higher score means better quality of life.
Biomarker of inflammation and exercise | From baseline to four months
  Difference in change in serum level Cathepsin-B (unit mikro gram/L)
MRI - Cerebral bloodflow | From baseline to four months
  Change in cerebral blood flow measured with arterial spin labeling (ASL) during rest
fMRI - Effective connectivity | From baseline to four months
  Change in activation patterns measured with blood-oxygen-level dependent (BOLD) during both single and bimanual task.
fMRI - Interhemispheric inhibition | From baseline to four months
  Change in activation pattern measured by blood-oxygen-level dependent (BOLD) during both single and bimanual task.
fMRI - Laterality Index | From baseline to four months
  Change in activation pattern for hemispheric dominance measured by the ratio of active fMRI voxels in each hemisphere.
MRI - Corticospinal integrity | From baseline to four months
  Change in corticospinal integrity measured by diffusion MRI.
MRI - Infarct lesion load | From baseline to four months
  Difference in change in size of infarct lesion meaured by structural MRI.
Upper-extremity motor outcome | From baseline to four months
  Follow-up Upper-extremity Fugl-Meyer Assessment (UE-FMA) score adjusted for baseline. Range 0-66
Feasibility: TDCS sensations | During intervention
  Proportion of participants experiencing sensations of TDCS (itching, pain, burning, vertigo, headache, fatigue, nausea, and/or other)
Feasibility: Compliance to interventions | During intervention
  Proportion of TDCS-intervention sessions attended out of the 12 planned sessions
Feasibilitiy: Compliance to home-exercises | During intervention
  Extent to which the participant has completed the planned home exercises ('fully', 'most', 'about 50%', 'below 50%', or 'not done')
Feasibility: Patient feed-back | Follow-up1
  The patients are asked if they would recommend TDCS to a peer patient (Yes/No)

OTHER OUTCOMES:
Brain Derived Neutrotrophic Factor (BDNF) genetic polymorphism | Baseline
  Determination of BDNF genetic variant - either Val66Met variant or wildtype.
Feasibility of intervention | From baseline to four months
  Completion of intervention in the active vs. control group
TMS - motor evoked potential | Baseline
  Determination of existence of a MEP-response by TMS as an indicator of cortico-spinal tract integrity. Prognostic marker of motor recovery.
TMS - Ipsilateral silent period (iSP) | Baseline
  Determination of degree of interhemispheric inhibition unaffected vs. affected hemisphere
TMS - Short latency intracortical inhibition (SICI) | Baseline
  Determination of degree of interhemispheric inhibition unaffected vs. affected hemisphere
TMS - cortico-motor conduction time (CMCT) | Baseline
  Determination of conduction time from stimulation of cortical neurons to response measured in a peripheral muscle (FDI)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kruuse, MD, Prof, Principal Investigator — Herlev Gentofte Hospital, Department of Neurology
Locations (3):
- Denmark (3):
  - Copenhagen University Department of Nutrition and Exercise, Copenhagen
  - Department of Neurology, Herlev Gentofte Hospital, Herlev
  - Danish Research Centre for Magnetic Resonance, Hvidovre

IPD SHARING:
Plan to Share IPD: Yes
IPD can be accessed upon reasonable request and after evaluation from the investigator.